CLINICAL TRIAL: NCT00595309
Title: Effect of a Booster Dose of the Japanese Encephalitis Vaccine IC51 on Long Term Immunogenicity. An Uncontrolled, Open-label Phase 3 Study.
Brief Title: Effect of a Booster Dose of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IC51-311
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Biological: IC51

INTERVENTIONS:
Biological: IC51 — IC51, 6 mcg, intramuscular (i.m.) booster vaccination 15 months after the primary immunization

SUMMARY:
The objective is to assess the effect of a booster vaccination on immunogenicity of IC51 in terms of seroconversion rate.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy adults who completed the primary immunization in study IC51 309
* Male and female healthy subjects aged at least 18 years with written informed consent and either no childbearing potential or negative pregnancy test

Main Exclusion Criteria:

• History of immunodeficiency or immunosuppressive therapy, known Human Immunodeficiency Virus (HIV), or drug addiction including alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Eder, Study Director — Valneva Austria GmbH
Locations (3):
- Austria (2):
  - Medizinische Universität Wien, Universitätsklinik für Klinische Pharmakologie, Vienna
  - Zentrum für Reisemedizin, Dependance für klinische Studien, Vienna
- Berliner Zentrum Reise- und Tropenmedizin, Berlin, Germany

REFERENCES:
- [Derived] Eder S, Dubischar-Kastner K, Firbas C, Jelinek T, Jilma B, Kaltenboeck A, Knappik M, Kollaritsch H, Kundi M, Paulke-Korinek M, Schuller E, Klade CS. Long term immunity following a booster dose of the inactivated Japanese Encephalitis vaccine IXIARO(R), IC51. Vaccine. 2011 Mar 21;29(14):2607-12. doi: 10.1016/j.vaccine.2011.01.058. Epub 2011 Feb 1. PMID 21288804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects participating in preceeding study IC51-309 were contacted. First Subject In December 2007, Last Subject In March 2008; study sites: center of pharmacology and travel clinics
Pre-assignment Details: subjects participating in study IC51-309 without major Protocol Deviations
Groups:
- IC51 Booster Group: IC51, 6 mcg, intramuscular (i.m.) booster vaccination 15 months after the primary immunization in study IC51-309
Period: Overall Study
Arm/Group | IC51 Booster Group
Started | 198
Completed | 194
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — planned vaccination against yellow fever | 1
Not completed — acute infection after V0 | 1
Not completed — personal reason | 1

BASELINE CHARACTERISTICS:
Arm/Group | IC51 Booster Group
Number analyzed (Participants) | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 197
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 94
Region of Enrollment [Number; unit: participants]
  Austria | 103
  Germany | 95

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate
Time Frame: at Month 12 after booster
Population: Intent-To-Treat Population which includes all subjects entered into the study who received the booster vaccination
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | IC51 Booster Group
Number analyzed (Participants) | 198
percent | 98.5 [95.6 to 99.5]

2. Secondary Outcome: Safety and Adverse Events
Time Frame: up to Month 12 after booster
Reporting Status: Not Posted

3. Secondary Outcome: Seroconversion
Time Frame: at D28 and Month 6 after booster
Reporting Status: Not Posted

4. Secondary Outcome: Geometric Mean Titer
Time Frame: D28, Month 6 and Month 12 after booster
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IC51 Booster Group
Serious Adverse Events (participants affected / at risk) | 8/198
Other Adverse Events (participants affected / at risk) | 96/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC51 Booster Group (N=198)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1)
Breast Cosmetic Surgery (Surgical and medical procedures) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Booster Group (N=198)
Fatigue (General disorders) | 14
Influenza Like Illnes (General disorders) | 19
Nasopharyngitis (Infections and infestations) | 30
Headache (Nervous system disorders) | 22
Hypochronic Anaemia (Blood and lymphatic system disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Pyrexia (General disorders) | 5
Allergy To Animal (Immune system disorders) | 2
Acute Tonsillitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 7
Cystitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 6
Influenza (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Limb Injury (Injury, poisoning and procedural complications) | 2
Alanine Aminotransferase Increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other